CLINICAL TRIAL: NCT04961008
Title: Safety and Sustainability in Bottle PEP in Cystic Fibrosis
Brief Title: Bottle PEP in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2019. 424
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bottle-PEP (Experimental): Bottle-PEP
  Interventions: Other: Bottle-PEP
- Routine physiotherapy (Active Comparator): v
  Interventions: Other: Routine physiotherapy

INTERVENTIONS:
Other: Bottle-PEP — A device that gives positive pressure from a bottle with the help of a non deflating tube
  Arms: Bottle-PEP
Other: Routine physiotherapy — Routine pulmonary physiotherapy
  Arms: Routine physiotherapy

SUMMARY:
The study aims to investigate the sustainability of Bottle-PEP in patients with cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Acute exacerbation

Exclusion Criteria:

* Any contraindication using the Bottle - PEP such as the presence of pneumothorax

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | every 3 months
  distance of meters walked in 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided